CLINICAL TRIAL: NCT03314909
Title: The Efficacy of Initial Hemopurification Strategy for Acute Paraquat Poisoning in Adults: Study Protocol for a Randomized Controlled Trial (HeSAPP)
Brief Title: Initial Hemopurification Strategy for Acute Paraquat Poisoning in Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other); National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Yi Li, MD, Chief physician of Emergency Department, professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HeSAPP
Record Dates: First submitted 2017-10-10; First posted 2017-10-19 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Poisoning
Keywords: Renal Dialysis; Hemoperfusion; Paraquat
MeSH Terms: conditions — Poisoning | interventions — Renal Dialysis; Hemoperfusion

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Masking Description: This study is designed as a non-blinded trial because of the apparently different equipment of the interventions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hemodialysis (HD) (Experimental): Patients in this group would receive hemodialysis for 3 days consecutively besides conservative therapy.
  Interventions: Procedure: Hemodialysis
- Hemoperfusion (HP) (Experimental): Patients in this group would receive hemoperfusion for 3 days consecutively besides conservative therapy.
  Interventions: Procedure: Hemoperfusion
- HP-HD (Experimental): Patients in this group would receive hemoperfusion and hemodialysis concurrent therapy for 3 days consecutively besides conservative therapy.
  Interventions: Procedure: HP-HD
- Conservative (No Intervention): Patients in this group would receive basic supportive treatment, gastric lavage, glucosteroid and immunosuppressive drugs without any hemopurification.

INTERVENTIONS:
Procedure: Hemodialysis — Participants in this group will be catheterize in the internal jugular vein and connect to a hemodialysis machine.
  Arms: Hemodialysis (HD)
Procedure: Hemoperfusion — Participants in this group will be catheterize in the internal jugular vein and connect to a hemoperfusion machine.
  Arms: Hemoperfusion (HP)
Procedure: HP-HD — Participants in this group will be catheterize in the internal jugular vein and connect to a hemoperfusion machine and then a hemodialysis machine for one course.
  Arms: HP-HD

SUMMARY:
HeSAPP is a single-center, non-blinded, parallel-group randomized controlled trial studying the hemopurification strategy for acute paraquat(PQ) poisoned patients. The intervention to be investigated include hemodialysis (HD), hemoperfusion (HP), combined hemoperfusion-hemodialysis concurrent therapy (HP-HD) and conservative therapy. The object of the present trial is to investigate whether hemopurification therapy can reduce mortality compared with conservative therapy.

DETAILED DESCRIPTION:
Patients diagnosed with acute paraquat poisoning in the Emergency Room of the First Affiliated Hospital of Zhengzhou University would be stratified according to their urine dithionite test results and randomly assigned to four different groups: HD, HP, HP-HD and control (conservative therapy) group for different treatment. Arterial blood gas test, complete blood count, coagulation function, liver function, pancreatic function, urine dithionite test, renal function and chest radiographs would be closely monitored during treatment. Primary endpoint is 28-day mortality. Secondary endpoints include (1) survival time (from the time of PQ ingestion to the time of death), all-cause mortality at the 3rd, 7th and 60th day; (2) rate of necessary oxygen uptake and rate of mechanical ventilation; (3) in-hospital length of stay and ICU length of stay; (4) APACHE II score and PSS score; (5) rate of general complications, such as respiratory failure, acute kidney injury (AKI), acute liver failure, pancreas function abnormality and Multiple Organ Failure (MOF); (6) rate of intervention related complications, such as catheter placement related complications, thrombocytopenia and deep venous thrombosis; (7) rate of adverse events, which include unexpected death, severe hemorrhage or edema, unplanned extubation, coagulation in the extracorporeal circulation, blockage of cartridge, incorrect pipe connection, etc.

ELIGIBILITY:
Inclusion Criteria:

* Suspected paraquat ingestion history (intended or accidental), which is confirmed by positive urine dithionite result (light blue, navy blue and dark blue).
* Arriving at the ER within 24 hours after PQ digestion.
* No known current pregnancy or lactation.
* Absence of cardiac arrest after poisoning, and no previous or present history of chronic kidney disease, chronic liver disease, respiratory failure, COPD, asthma, heart failure, pancreatic disease, acute coronary syndrome (ACS) or stoke.
* No known combined ingestion with other poisons or alcohol.
* No previous blood purification treatment prior to admission.
* No known participation in other medical trials.
* Agreement on informed consent.

Exclusion Criteria:

* Patients who are unable to comply with the procedures of the present trial, including those who change therapy or withdraw treatment.
* Patients who develop severe allergic response to HP materials.
* Patients who do not receive intervention within 4 hours after admission in reality.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
28-day all-cause mortality | From the day of intoxication to the 28th day afterwards.
  Mortality=Dead patients/All patients in that group

SECONDARY OUTCOMES:
Survival time | From the day of intoxication to death or the 60th day.
  Live day count.
Rate of multiple organ failure | From the day of intoxication to death or the 60th day.
  Patients that develop multiple organ failure/All patients in that group
Rate of oxygen uptake | From the day of intoxication to death or the 60th day.
  Patients that need oxygen therapy/All patients in that group
Rate of mechanical ventilation | From the day of intoxication to death or the 60th day.
  Patients that need mechanical ventilation/All patients in that group
In-hospital length of stay | From the day of admission to discharge or up to 60 days after admission.
  Day count from admission to discharge or the end of follow up.
3-day all-cause mortality | From the day of intoxication to the 3rd day afterwards.
  Mortality=Dead patients/All patients in that group
7-day all-cause mortality | From the day of intoxication to the 7th day afterwards.
  Mortality=Dead patients/All patients in that group
60-day all-cause mortality | From the day of intoxication to the 60th day afterwards.
  Mortality=Dead patients/All patients in that group
ICU length of stay | From the day of intoxication to death or the 60th day.
  Day count spent in intensive care unit
Rate of catheter related complications | From the day of intoxication to death or the 60th day.
  Complications due to catheterization, e.g. thrombocytopenia, deep venous thrombosis, catheter related infection.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Li, M.D., Study Chair — Peking Union Medical College Hospital; Yanxia Gao, Study Director — The First Affiliated Hospital of Zhengzhou University

IPD SHARING:
Plan to Share IPD: Undecided
Not decided.

REFERENCES:
- [Derived] Cui JW, Xu Y, Wang Y, Gao YX, Guo S, Wang M, Lu X, Yu S, Ma Y, Yuan D, Che L, Sun P, Yu X, Zhu H, Li Y. Efficacy of initial haemopurification strategy for acute paraquat poisoning in adults: study protocol for a randomised controlled trial (HeSAPP). BMJ Open. 2018 Jun 22;8(6):e021964. doi: 10.1136/bmjopen-2018-021964. PMID 29934393

DOCUMENTS (2):
  • Study Protocol (2018-04-06): https://cdn.clinicaltrials.gov/large-docs/09/NCT03314909/Prot_002.pdf
  • Statistical Analysis Plan (2018-04-06): https://cdn.clinicaltrials.gov/large-docs/09/NCT03314909/SAP_003.pdf